CLINICAL TRIAL: NCT00001770
Title: The Phenomenology and Biophysiology of Progestin-Induced Dysphoria
Brief Title: Progestin (Progesterone-Like Hormones) Induced Dysphoria (Depressed Mood, Irritability, Anxiety)
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980079; 98-M-0079
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-03

CONDITIONS: Depressive Disorder; Mood Disorder; Psychomotor Agitation
Keywords: Depression; Estrogen; Hormone Replacement Therapy; Mood; Progestin; Progesterone; Anxiety
MeSH Terms: conditions — Depressive Disorder; Mood Disorders; Psychomotor Agitation; Depression; Anxiety Disorders

SUMMARY:
Often women are prescribed hormone replacement therapy (HRT) during the perimenopause or menopause.

Hormone replacement therapy includes both estrogen and progesterone. The estrogen component of HRT helps to relieve the symptoms and has a beneficial effect on the heart and bones, but estrogen also increases the risk of uterine cancer. The progesterone component of the HRT (progestin) works to prevent the increased risk of uterine cancer.

There is evidence that some women experience unpleasant mood symptoms (such as irritability, depressed mood and anxiety) while receiving hormone replacement therapy (HRT) while taking the progestin / progesterone component of the HRT.

This study is designed to evaluate the ability of progestins to produce negative mood symptoms in women. Researchers intend on doing this by comparing the effects of medroxyprogesterone acetate (Provera) and a placebo inactive sugar pill. Patient's moods will be monitered based on their response to questionnaires answered in the outpatient clinic and at home.

This research will attempt to answer the following questions:

1. Are progestins associated with changes in mood during hormone replacement therapy?
2. If progestins are associated with mood disturbance, is it because they are blocking the beneficial effects of estrogen?

DETAILED DESCRIPTION:
There is evidence in the literature that some women experience dysphoric symptoms while receiving hormone replacement therapy (HRT) and that this disturbance in mood is related to the progestin component of the HRT. The bulk of this evidence is anecdotal. While some authors have attempted to examine this putative problem in a more systematic fashion, there are no controlled studies that attempt to identify the mechanism through which the perturbation in mood occurs. Adverse effects of progestins might be mediated directly through the progesterone or androgen receptor. Alternatively, the effects of progestins might be consequent to the antiestrogen effects of progesterone. This latter possibility is in part supported by our observation in previous studies of the beneficial effects of estradiol on mood and the possible precipitation of mood disturbance following acute estrogen withdrawal. Finally, despite the popular lore that progesterone causes mood disturbances, a placebo effect cannot be ruled out, since women taking HRT know when they are receiving the progestin component of the regimen. Our research questions therefore are as follows: 1) Are progestins associated with changes in mood during HRT, and 2) If progestins are associated with mood disturbance, is it because they are blocking the beneficial effects of estrogen?

ELIGIBILITY:
INCLUSION CRITERIA

The subjects in this study will be women who meet the following criteria:

1. history of mood and/or behavioral symptoms associated with hormone replacement therapy;
2. age 40 to 65;
3. in good medical health.

EXCLUSION CRITERIA

Any subject with significant physical, EKG, mammogram or laboratory abnormalities will not participate in this protocol. Additionally prior to participation all subjects will be examined for any contradictions to estrogen therapy (as determined by a pelvic exam and mammogram) within the past year by a gynecologist of their choice. In those patients who are unable to independently arrange this exam, we have arranged for a consultant gynecologist to be available through our collaboration with NICHD.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1998-03; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Wagner KD. Major depression and anxiety disorders associated with Norplant. J Clin Psychiatry. 1996 Apr;57(4):152-7. PMID 8601550
- [Background] Smith RN, Holland EF, Studd JW. The symptomatology of progestogen intolerance. Maturitas. 1994 Feb;18(2):87-91. doi: 10.1016/0378-5122(94)90046-9. PMID 8177097
- [Background] Magos AL, Brewster E, Singh R, O'Dowd T, Brincat M, Studd JW. The effects of norethisterone in postmenopausal women on oestrogen replacement therapy: a model for the premenstrual syndrome. Br J Obstet Gynaecol. 1986 Dec;93(12):1290-6. doi: 10.1111/j.1471-0528.1986.tb07868.x. PMID 3801360